CLINICAL TRIAL: NCT06244680
Title: Super-fast 3T Prostate MRI Using High Gradient Strength and Deep Learning: Initial Experience
Brief Title: Super-fast 3T Prostate MRI Using High Gradient Strength and Deep Learning
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, PD Dr. med.; Head of MR-Imaging, University Hospital, Bonn
Other Study IDs: CX.001
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MRI of the prostate — Patients with suspicion for prostate cancer underwent mpMRI on a new 3-Tesla-MRI scanner with a maximum gradient strength of 200 mT/m, a slew rate of 200 T/m/s and DL reconstruction for image postprocessing.

SUMMARY:
Recent developments in MRI techniques allow ultra-high gradient strength diffusion imaging and deep learning (DL) reconstruction in clinical routine. However, its usability in biparametric MRI (bpMRI) of the prostate has not been well studied. The aim is to establish a super-fast 3-minutes bpMRI protocol at 3 Tesla using high gradient strength and DL reconstruction and compare it against a full, multiparametric MRI (mpMRI) protocol.

DETAILED DESCRIPTION:
Multiparametric MRI (mpMRI) of the prostate has become the most important non-invasive diagnostic tool for assessment of prostate cancer and is the baseline for MRI targeted biopsy (1,2). As the incidence of prostate cancer is high with an estimated 290,000 new cases for 2023 in the United States alone (3), the need for widespread provision of prostate mpMRI is immense. However, current clinical MRI-protocols are long with acquisition times of >30 minutes, potentially limiting the number of examined patients. According to the guidelines of the Prostate Imaging Reporting and Data System (PI-RADS) a sufficient mpMRI protocol must include diffusion weighted imaging (DWI), T2-weighted (T2w) imaging, dynamic contrast enhanced imaging and T1-weighted imaging pre and post administration of contrast (4,5). Different approaches have been developed to shorten the protocol itself or to accelerate acquisition times. For instance, a significant reduction of T2w-sequence acquisition times was achieved by employing deep learning methods (6) or advancements of compressed sensing (7), while at the same time images had improved quality. Different studies showed equal performance of biparametric MRI (bpMRI) protocols compared to the standard multiparametric protocol, effectively reducing the acquisition time down to 5 minutes (8,9,10). This was done by focusing only on DWI and T2w imaging while omitting the dynamic contrast enhanced sequence and T1-weighted sequences, as the additional diagnostic value of these is supposed to be limited (11).

Recent developments in MRI techniques allow for ultra-high diffusion gradient strengths of up to 500 mT/m and slew rates of up to 600 T/m/s, thus reducing echo times and acquisition times by faster establishment of the diffusion gradient (12,13). Furthermore, these gradients are able to image at small scales with a high signal-to-noise ratio, consecutively enhancing sensitivity for detection of tissue microstructures (14,15). Due to the experimental nature of these gradients, this technique has only been investigated in a research setting in healthy volunteers (16), but not in a real world clinical setting, let alone in prostate imaging.

Therefore, the aim of the study was to establish a super-fast abbreviated bpMRI protocol for patients with suspicion for prostate cancer using both ultra-high gradients and deep learning reconstruction for DWI- and T2w-sequences. Besides the assessment of acquisition times, the main objective of this study was to assess the overall image quality of bpMRI and mpMRI and the influence on PI-RADS scores.

ELIGIBILITY:
Inclusion Criteria:

* Elevated PSA >4ng/ml or suspicious digitial rectal exam or supicious transrectal ultrasound

Exclusion Criteria:

* General MRI contraindications (incompatible cardiac pacemaker, neurostimulators) or allergy for gadolinium-containing contrast media or severe claustrophobie

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of male patients with clinical suspicion for prostate cancer, as described by the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Agreement of PI-RADS scores | January - February 2024
  Three radiologists with 3, 11 and 12 years of experience in prostate MRI read separately and blinded to personal and clinical parameters (name, age, patient history, value of the prostate specific antigen, clinical examination and transrectal ultrasound) the full bpMRI protocol and graded the lesions according to the PI-RADS classification. Per patient, only the highest graded lesion and its respective prostate zone was noted. If there were two distinct lesions with the highest PI-RADS score in both the peripheral and transitional zone, both were noted. After a washout period of one month all readers did the same for the mpMRI protocol. Both the agreement of biparametric and multiparametric MRI PI-RADS scores for the whole prostate, and for the specific zonal distribution (peripheral and transitional zone) were assessed by calculation of Cohens's κ, interpreted as follows: <0.5 = poor; 0.5-0.75 = moderate; 0.75-0.9 = good; >0.9 = excellent.
Acquisition time | January - February 2024
  Acquisition times for the whole biparametric and whole multiparametric protocol was measured.
Image quality | January - February 2024
  Two raters with 3 and 11 years of experience rated the bpMRI protocol on a five point Likert scale in six different qualitative categories (artifacts, image sharpness, lesion conspicuity, capsule delineation, overall image sharpness and diagnostic confidence). The grades were defined as follows: 1, non-diagnostic due to extensive artifacts, strongly impaired conspicuity of anatomical structures and no diagnostic confidence; 2, several artifacts, difficult conspicuity of anatomical structures and low diagnostic confidence; 3, moderate artifacts, fair conspicuity of anatomical structures and moderate diagnostic confidence; 4, little artifacts, good conspicuity of anatomical structures and good diagnostic confidence; 5, no artifacts, excellent conspicuity of anatomical structures and high diagnostic confidence. Results of both raters were averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Julian A Luetkens, PD Dr. med, Principal Investigator — University of Bonn
Locations (1):
- University Hospital Bonn, Clinic for Diagnostic and Interventional Radiology, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hugosson J, Mansson M, Wallstrom J, Axcrona U, Carlsson SV, Egevad L, Geterud K, Khatami A, Kohestani K, Pihl CG, Socratous A, Stranne J, Godtman RA, Hellstrom M; GOTEBORG-2 Trial Investigators. Prostate Cancer Screening with PSA and MRI Followed by Targeted Biopsy Only. N Engl J Med. 2022 Dec 8;387(23):2126-2137. doi: 10.1056/NEJMoa2209454. PMID 36477032
- [Background] Eklund M, Jaderling F, Discacciati A, Bergman M, Annerstedt M, Aly M, Glaessgen A, Carlsson S, Gronberg H, Nordstrom T; STHLM3 consortium. MRI-Targeted or Standard Biopsy in Prostate Cancer Screening. N Engl J Med. 2021 Sep 2;385(10):908-920. doi: 10.1056/NEJMoa2100852. Epub 2021 Jul 9. PMID 34237810
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] ACR, ESUR and AdMeTech Foundation. Prostate Imaging Reporting & Data System (PI-RADS). 2019. Version 2.1.
- [Background] Hegde JV, Mulkern RV, Panych LP, Fennessy FM, Fedorov A, Maier SE, Tempany CM. Multiparametric MRI of prostate cancer: an update on state-of-the-art techniques and their performance in detecting and localizing prostate cancer. J Magn Reson Imaging. 2013 May;37(5):1035-54. doi: 10.1002/jmri.23860. PMID 23606141
- [Background] Bischoff LM, Peeters JM, Weinhold L, Krausewitz P, Ellinger J, Katemann C, Isaak A, Weber OM, Kuetting D, Attenberger U, Pieper CC, Sprinkart AM, Luetkens JA. Deep Learning Super-Resolution Reconstruction for Fast and Motion-Robust T2-weighted Prostate MRI. Radiology. 2023 Sep;308(3):e230427. doi: 10.1148/radiol.230427. PMID 37750774
- [Background] Bischoff LM, Katemann C, Isaak A, Mesropyan N, Wichtmann B, Kravchenko D, Endler C, Kuetting D, Pieper CC, Ellinger J, Weber O, Attenberger U, Luetkens JA. T2 Turbo Spin Echo With Compressed Sensing and Propeller Acquisition (Sampling k-Space by Utilizing Rotating Blades) for Fast and Motion Robust Prostate MRI: Comparison With Conventional Acquisition. Invest Radiol. 2023 Mar 1;58(3):209-215. doi: 10.1097/RLI.0000000000000923. Epub 2022 Sep 2. PMID 36070533
- [Background] Weiss J, Martirosian P, Notohamiprodjo M, Kaufmann S, Othman AE, Grosse U, Nikolaou K, Gatidis S. Implementation of a 5-Minute Magnetic Resonance Imaging Screening Protocol for Prostate Cancer in Men With Elevated Prostate-Specific Antigen Before Biopsy. Invest Radiol. 2018 Mar;53(3):186-190. doi: 10.1097/RLI.0000000000000427. PMID 29077588
- [Background] Scialpi M, Prosperi E, D'Andrea A, Martorana E, Malaspina C, Palumbo B, Orlandi A, Falcone G, Milizia M, Mearini L, Aisa MC, Scialpi P, DE Dominicis C, Bianchi G, Sidoni A. Biparametric versus Multiparametric MRI with Non-endorectal Coil at 3T in the Detection and Localization of Prostate Cancer. Anticancer Res. 2017 Mar;37(3):1263-1271. doi: 10.21873/anticanres.11443. PMID 28314291
- [Background] Rais-Bahrami S, Siddiqui MM, Vourganti S, Turkbey B, Rastinehad AR, Stamatakis L, Truong H, Walton-Diaz A, Hoang AN, Nix JW, Merino MJ, Wood BJ, Simon RM, Choyke PL, Pinto PA. Diagnostic value of biparametric magnetic resonance imaging (MRI) as an adjunct to prostate-specific antigen (PSA)-based detection of prostate cancer in men without prior biopsies. BJU Int. 2015 Mar;115(3):381-8. doi: 10.1111/bju.12639. Epub 2014 Sep 15. PMID 24447678
- [Background] De Visschere P, Lumen N, Ost P, Decaestecker K, Pattyn E, Villeirs G. Dynamic contrast-enhanced imaging has limited added value over T2-weighted imaging and diffusion-weighted imaging when using PI-RADSv2 for diagnosis of clinically significant prostate cancer in patients with elevated PSA. Clin Radiol. 2017 Jan;72(1):23-32. doi: 10.1016/j.crad.2016.09.011. Epub 2016 Oct 7. PMID 27726850
- [Background] Huang SY, Witzel T, Keil B, Scholz A, Davids M, Dietz P, Rummert E, Ramb R, Kirsch JE, Yendiki A, Fan Q, Tian Q, Ramos-Llorden G, Lee HH, Nummenmaa A, Bilgic B, Setsompop K, Wang F, Avram AV, Komlosh M, Benjamini D, Magdoom KN, Pathak S, Schneider W, Novikov DS, Fieremans E, Tounekti S, Mekkaoui C, Augustinack J, Berger D, Shapson-Coe A, Lichtman J, Basser PJ, Wald LL, Rosen BR. Connectome 2.0: Developing the next-generation ultra-high gradient strength human MRI scanner for bridging studies of the micro-, meso- and macro-connectome. Neuroimage. 2021 Nov;243:118530. doi: 10.1016/j.neuroimage.2021.118530. Epub 2021 Aug 28. PMID 34464739
- [Background] Fan Q, Eichner C, Afzali M, Mueller L, Tax CMW, Davids M, Mahmutovic M, Keil B, Bilgic B, Setsompop K, Lee HH, Tian Q, Maffei C, Ramos-Llorden G, Nummenmaa A, Witzel T, Yendiki A, Song YQ, Huang CC, Lin CP, Weiskopf N, Anwander A, Jones DK, Rosen BR, Wald LL, Huang SY. Mapping the human connectome using diffusion MRI at 300 mT/m gradient strength: Methodological advances and scientific impact. Neuroimage. 2022 Jul 1;254:118958. doi: 10.1016/j.neuroimage.2022.118958. Epub 2022 Feb 23. PMID 35217204
- [Background] Setsompop K, Kimmlingen R, Eberlein E, Witzel T, Cohen-Adad J, McNab JA, Keil B, Tisdall MD, Hoecht P, Dietz P, Cauley SF, Tountcheva V, Matschl V, Lenz VH, Heberlein K, Potthast A, Thein H, Van Horn J, Toga A, Schmitt F, Lehne D, Rosen BR, Wedeen V, Wald LL. Pushing the limits of in vivo diffusion MRI for the Human Connectome Project. Neuroimage. 2013 Oct 15;80:220-33. doi: 10.1016/j.neuroimage.2013.05.078. Epub 2013 May 24. PMID 23707579
- [Background] McNab JA, Edlow BL, Witzel T, Huang SY, Bhat H, Heberlein K, Feiweier T, Liu K, Keil B, Cohen-Adad J, Tisdall MD, Folkerth RD, Kinney HC, Wald LL. The Human Connectome Project and beyond: initial applications of 300 mT/m gradients. Neuroimage. 2013 Oct 15;80:234-45. doi: 10.1016/j.neuroimage.2013.05.074. Epub 2013 May 24. PMID 23711537
- [Background] Huang SY, Tian Q, Fan Q, Witzel T, Wichtmann B, McNab JA, Daniel Bireley J, Machado N, Klawiter EC, Mekkaoui C, Wald LL, Nummenmaa A. High-gradient diffusion MRI reveals distinct estimates of axon diameter index within different white matter tracts in the in vivo human brain. Brain Struct Funct. 2020 May;225(4):1277-1291. doi: 10.1007/s00429-019-01961-2. Epub 2019 Sep 28. PMID 31563995
- [Derived] Bischoff LM, Endler C, Krausewitz P, Ellinger J, Klumper N, Isaak A, Mesropyan N, Kravchenko D, Nowak S, Kuetting D, Sprinkart AM, Murtz P, Pieper CC, Attenberger U, Luetkens JA. Ultra-high gradient performance 3-Tesla MRI for super-fast and high-quality prostate imaging: initial experience. Insights Imaging. 2024 Nov 29;15(1):287. doi: 10.1186/s13244-024-01862-x. PMID 39614012